CLINICAL TRIAL: NCT02468830
Title: Prospective Pilot Study of Mirabegron in Pediatric Patients With Overactive Bladder
Brief Title: Pilot Study of Mirabegron in Pediatric Patients With Overactive Bladder
Acronym: Mirabegron
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Principal Investigator, Stéphane Bolduc, Pediatric Urologist, MD, FRCSC, FAAP, CHU de Quebec-Universite Laval
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B14-06-1998
Record Dates: First submitted 2015-05-30; First posted 2015-06-11 (Estimated); Results first posted 2018-06-20 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Overactive Bladder; Urinary Incontinence
Keywords: mirabegron; antimuscarinics; beta 3 agonist; overactive bladder; children
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence | interventions — mirabegron

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mirabegron (Experimental): Patients without symptom improvement or with partial response under intensive behavioural protocol and medical therapy (at least 2 different antimuscarinic agents) will be recruited. Patients with significantly bothersome S/E on antimuscarinics will also be included.
  Interventions: Drug: mirabegron

INTERVENTIONS:
Drug: mirabegron — Switch treatment from antimuscarinic to study medication. A dose up-titration will be possible if well tolerated and sub-optimal efficacy.
  Other Names: Myrbetriq

SUMMARY:
The objective is to evaluate the efficacy and safety of mirabegron to treat urinary incontinence in children with Overactive Bladder that are refractory and/or intolerant to antimuscarinics.

DETAILED DESCRIPTION:
Overactive bladder (OAB) is a highly prevalent disorder in the pediatric population. This condition comprises many urinary symptoms, such as urgency, increased daytime frequency of micturition, urge incontinence and nocturia. These symptoms are especially troublesome for the pediatric patients and their family since it causes embarrassment and it limits everyday activities and impairs children's development. Furthermore, serious complications are seen if this condition is not treated properly, as urinary tract infection, vesico-ureteral reflux and dysfunctional voiding. Antimuscarinic agents are the current pharmacologic mainstay for OAB. Many side effects are reported with the clinical use of antimuscarinics. Oxybutynin is the most widely antimuscarinic agent used in the pediatric population and is the only molecule approved by Health Canada for children with OAB. However, some patients have a suboptimal response to antimuscarinic and many experience side effects. Children with OAB therefore represent a disease population with a need for an alternative effective, safe and well-tolerated therapy to help manage the overactive detrusor, reducing or preventing incontinence.

Mirabegron, a β3-adrenoceptor (β3-AR) agonist approved for the treatment of OAB symptoms in the adult population, is the first of a new class of compounds with a different mechanism of action. The recommended starting dose of mirabegron is 25mg, which can be increased to 50mg, based on individual efficacy and tolerability. Side effects commonly reported with antimuscarinics were not observed more often with mirabegron than with placebo (headache 2.0%, dry mouth 2.0%, constipation 1.6%). Several Phase II and III studies have shown significant improvement in clinical OAB symptoms in adults treated with mirabegron with a favorable tolerability profile. Mirabegron has not been studied yet for pediatric patients and no recommendation with regards to its use has been issued by the manufacturer nor medical regulatory bodies.

A prospective open-label study, using an adjusted-dose regimen of mirabegron (25-50mg), including pediatric patients with refractory urinary incontinence due to OAB. This protocol was approved by the investigators' research ethics board. Patients without symptom improvement or with partial response under intensive behavioural protocol and medical therapy (at least 2 different antimuscarinic agents) will be recruited. Patients with significantly bothersome S/E on antimuscarinics are also included. primary end-point is efficacy toward urinary continence and secondary end-points are tolerability and safety. The patients/parents satisfaction will also be recorded.

After 8 to 12 weeks on the new medication, the possibility of up-titration will be assessed. Patients and parents will be questioned on compliance, tolerability and efficacy. If the patient is taking the medication ≥80% of the time, does not have any significant side effects and still has significant OAB symptoms, the investigators will offer a dose increase (Mirabegron 50mg daily). If accepted, the medication will be provided with instructions to report any new side effects.

Subjects will complete a 3-day voiding diary prior to each medical visit to assess the efficacy of the treatment and urotherapy. Visits will be done every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 5 years old and ≤17 years old
* OAB diagnostic according to the International Children Continence Society (ICCS) and less than 65% of the expected mean bladder capacity for age is confirmed (30 + (age in years x 30) mL) on a 3-day voiding diary.
* Weight and height are within the normal percentile (3rd to 97th percentile) and weight is ≥ 20 kg (3rd percentile of a 8 y.o. child, boy or girl), according to the CDC growth chart
* Ability to swallow pills
* Subjects/parents (vs. legal guardian) agree to participate to the following study and sign the informed consent
* Subjects/parents (vs. legal guardian) are able to comply with the study requirements and with the medication restrictions.
* Female subjects of childbearing potential must have a negative serum or urine pregnancy test at enrollment and must agree to maintain highly effective birth control during the study. Sexually active male subjects agree to use a barrier method of birth control with female partner for the duration of the study and at least one month after ending study treatment. Sexually active male subjects agree to use a condom for the duration of the study and for at least one month after ending study treatment and the female partner to use a reliable form of birth control for the duration of the study and for at least one month after ending study treatment.
* Patients without symptom improvement or with partial response under medical therapy (at least 2 different antimuscarinic agents) or with significantly bothersome S/E on antimuscarinics.

Exclusion Criteria:

* Subject has a diagnostic of dysfunctional voiding
* Post-voiding residue > 20 cc
* Polyuria (> 75 ml/kg/b.w./24 hours)
* Nephrogenic of central diabetes insipidus
* Constipation at screening (if the patient is treated and the treatment is successful, the patient will be eligible to the study)
* Urinary tract infection at visit 2-3-4. If UTI is present at the screening visit, the UTI must be treated and the success of the treatment must be documented with a negative urinalysis at visit 2.
* QTc interval greater than 460 ms, or any increase of 30 ms on follow-up EKG (mean of 6 separate EKG-3 from visit week-2 and 3 from visit week 0). If a patient meets those criteria in the first month (initial dose), he will be excluded from the study. If the QTc change is noted after the up-titration, the dose will be decreased and EKG will be repeated within 1 week to ensure normalization of QTc.
* Clinically significant unstable medical condition or disorder
* Subject is pregnant or intends to become pregnant
* Serum creatinin more than or equal to 2 times the upper limit of normal
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) more than or equal to 2 times ULN, or bilirubin more than or equal to 1.5 times ULN.
* Known hypersensitivity to mirabegron or any contraindication to the use of the molecule, in accordance to the product monography (to the exception of pediatric age).
* Subject is taking medication that interact with mirabegron and this medication can't be discontinued (see appendix 1 of excluded drugs)
* Known urological pathology other than OAB that could explain urinary symptoms (as bladder stone…)
* Non-treated or non-controlled arterial hypertension

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2013-04; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
Publication submitted
Supporting Information: CSR
Time Frame: March 2018
Access Criteria: publication

REFERENCES:
- [Result] Blais AS, Nadeau G, Moore K, Genois L, Bolduc S. Prospective Pilot Study of Mirabegron in Pediatric Patients with Overactive Bladder. Eur Urol. 2016 Jul;70(1):9-13. doi: 10.1016/j.eururo.2016.02.007. Epub 2016 Feb 11. PMID 26876327

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mirabegron
Started | 58
Completed | 55
Not Completed | 3

BASELINE CHARACTERISTICS:
Groups:
- Mirabegron: Patients without symptom improvement or with partial response under intensive behavioural protocol and medical therapy (at least 2 different antimuscarinic agents) will be recruited. Patients with significantly bothersome S/E on antimuscarinics will also be included.
  mirabegron (initial dosage 25 mg this dose wil be maintain or increase to a maximum of 50 mg based on persistent of symptomsand side effect profile): Switch treatment from antimuscarinic to study medication. A dose up-titration will be possible if well tolerated and sub-optimal efficacy.
Arm/Group | Mirabegron
Number analyzed (Participants) | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 58
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 44
Region of Enrollment [Number; unit: participants]
  Canada | 58

OUTCOME MEASURES:

1. Primary Outcome: Improved Overactive Bladder Symptoms as a Measure of Efficacy of Mirabegron
Description: Percent change in the frequency of urinary incontinence episodes as a Measure of Efficacy.
Time Frame: Participants will be followed for the duration of the study, up to 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Mirabegron
Number analyzed (Participants) | 58
Participants
  Complete elimination of urinary incontinence:100% | 13
  Significant response > 90%- | 14
  Partial response: 50-89% | 25
  Failure < 50% | 6

2. Primary Outcome: Improved Overactive Bladder Symptoms as a Measure of Efficacy of Mirabegron
Description: Change in mean bladder capacity from baseline to final visit based on voiding diary.
Time Frame: Participants will be followed for duration of the study, up to 52 weeks
Measure: Median (Inter-Quartile Range); unit: milliliter
Arm/Group | Mirabegron
Number analyzed (Participants) | 58
milliliter
  baseline | 150 [125 to 200]
  Final visit | 200 [171 to 300]

3. Secondary Outcome: Number of Participants With Cardio Vascular Safety
Description: Cardiovascular safety: mean difference in blood pressure (Variation in blood pressure: systolic ±20 mmHg, diastolic ±15 mmHg).
  Parameters to be measure at each visit but particularly at visit 2 (Week 0, first dose on site), to be obtained before and 1 hour after taking the medication).
Time Frame: Participants will be followed for the duration of the study, up to 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Mirabegron
Number analyzed (Participants) | 58
Participants
  No variation:systolic ±20 mmHg in blood pressure | 58
  No variation:Diastolic ±15 mmHg in blood pressure | 58

4. Secondary Outcome: Improved Quality of Life Using the Patient Perception of Bladder Condition (PPBC) Scale
Description: The Patient Perception of Bladder Condition (PPBC) scale on a 6-point score scale at baseline and final visit.
  Explanation of possible answer:
  1. does not cause me any problems at all,
  2. causes me some very minor problems,
  3. causes me some minor problems,
  4. causes me (some) moderate problems,
  5. causes me severe problems,
  6. causes me many severe problems
Time Frame: Participants will be followed for the duration of the study, up to 52 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Mirabegron
Number analyzed (Participants) | 58
units on a scale
  baseline | 4.0 [4.0 to 5.0]
  Final visit | 2.0 [1.0 to 3.0]

5. Secondary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability of Mirabegron
Description: Cardiovascular safety: mean difference in heart rate (variation in heart rate increase of more than 20%). Heart rate was taken at initiation of study drug, at each visit and at the study end.
Time Frame: Participants will be followed for the duration of the study, up to 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Mirabegron
Number analyzed (Participants) | 58
Participants
  No change in heart rate over 20% | 58
  No significant change in heart rate | 58

ADVERSE EVENTS:
Arm/Group | Mirabegron
Serious Adverse Events (participants affected / at risk) | 0/58
Other Adverse Events (participants affected / at risk) | 8/58
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mirabegron (N=58)
Transient abdominal colic (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Blurred vision (Eye disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Change in behavior (General disorders) | 1 (1)
Nasopharyngitis (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No